CLINICAL TRIAL: NCT02499510
Title: First-in-man Study to Assess Efficacy and Safety of a Novel Titanium-Nitride Coated Woven-nitinol Peripheral Arterial Stent
Brief Title: First-in-man Study of Titanium-Nitride Coated Woven-nitinol Peripheral Arterial Stent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Lifetech Scientific (Shenzhen) Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Professor Bryan Ping Yen YAN, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Not_applicable
Record Dates: First submitted 2015-05-11; First posted 2015-07-16 (Estimated); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Peripheral Arterial Disease
Keywords: femoropopliteal disease; restenosis
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GoldenFlow stent (Experimental): Titanium nitrite coated woven nitinol stent
  Interventions: Device: GoldenFlow Stent

INTERVENTIONS:
Device: GoldenFlow Stent — The GoldenFlow stent (Lifetech Science, Shenzhen, China) is a TiN coated self-expanding stent consisting of interwoven nitinol wires braided in a closed cell design. Stents used in this study ranged from 4-12mm in diameter and 20-160mm in length.
  Other Names: Titanium-nitride coated GoldenFlow woven-nitinol stent

SUMMARY:
The GoldenFlow (Lifetech Scientific, Shenzhen, China) is a novel woven-nitinol stent designed to have superior radial strength, flexibility and durability compared to standard nitinol stents for femoropopliteal lesions. This is a first-in-man study to evaluate the safety and efficacy of GoldenFlow woven-nitinol stent for intraluminal treatment of peripheral vascular disease in the femoropopliteal arteries.

DETAILED DESCRIPTION:
Endovascular treatment in femoropopliteal segment is the most challenging area due to restenosis and stent fracture after endovascular treatment. The titanium-nitride coated woven-nitinol peripheral arterial stent system (GoldenFlow, Lifetech Science, Shenzhen, China) is designed to have superior radial strength, flexibility and durability to withstand the compression, torsion, bending, lengthening and shortening found in femoropopliteal disease. Compared to another commercially available woven-nitinol stent, the GoldenFlow stent has the potential advantage to be repositionable and is less likely to lengthen during deployment. This is a first-in-man study is to evaluate the safety and efficacy of GoldenFlow woven-nitinol stent for intraluminal treatment of peripheral vascular disease in de-novo femoropopliteal lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Symptomatic leg ischemia (Rutherford class 2 to 4)
3. Ankle Brachial Index <0.9
4. De novo femoropopliteal stenosis (≥70%) or occlusion
5. Reference diameter 4 and 7mm
6. Lesion length 4 to 15cm
7. At least one patent (<50% stenosis) infrapopliteal run-off vessel
8. The lesion(s) can be successfully crossed with a guidewire and dilated
9. Patients with bilateral femoropopliteal disease is eligible for enrollment into the study

   - Staged contralateral limb procedure can be performed >30 days after index procedure
10. Able to provide written informed consent and willing to comply with specified follow-up evaluation schedule

Exclusion Criteria:

1. Tissue loss or gangrene (Rutherford class 5 and 6)
2. Previous bypass surgery or stenting in target vessel
3. Untreated aortoiliac or common femoral artery inflow disease >50%
4. Intervention of ipsilateral lesions during the index procedure or staged intervention within 30 days after index procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-10; Primary Completion 2017-11 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
In-stent binary restenosis of the treated segment | at 6 month
  Determined by Duplex ultrasound

SECONDARY OUTCOMES:
Technical Success | intraoperation
  defined as residual diameter stenosis <30%
Safety Outcomes as assessed by composite of death, index limb amputation and ischemic driven target vessel revacularization | 30 days
  Composite of death, index limb amputation and ischemic driven target vessel revacularization at 30 days
Clinically driven target vessel revascularization | 6 months
Stent fracture | 6 months
  defined by plain x-ray

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Ping Yen Yan, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, New Territories, Hong Kong

REFERENCES:
- [Background] Dormandy JA, Rutherford RB. Management of peripheral arterial disease (PAD). TASC Working Group. TransAtlantic Inter-Society Consensus (TASC). J Vasc Surg. 2000 Jan;31(1 Pt 2):S1-S296. No abstract available. PMID 10666287
- [Background] Johnston KW. Femoral and popliteal arteries: reanalysis of results of balloon angioplasty. Radiology. 1992 Jun;183(3):767-71. doi: 10.1148/radiology.183.3.1294068.
- [Background] Minar E, Pokrajac B, Maca T, Ahmadi R, Fellner C, Mittlbock M, Seitz W, Wolfram R, Potter R. Endovascular brachytherapy for prophylaxis of restenosis after femoropopliteal angioplasty : results of a prospective randomized study. Circulation. 2000 Nov 28;102(22):2694-9. doi: 10.1161/01.cir.102.22.2694. PMID 11094034
- [Background] Capek P, McLean GK, Berkowitz HD. Femoropopliteal angioplasty. Factors influencing long-term success. Circulation. 1991 Feb;83(2 Suppl):I70-80. PMID 1825050
- [Background] Henry M, Amor M, Beyar R, Henry I, Porte JM, Mentre B, Tricoche O, Ethevenot G. Clinical experience with a new nitinol self-expanding stent in peripheral arteries. J Endovasc Surg. 1996 Nov;3(4):369-79. doi: 10.1583/1074-6218(1996)0032.0.CO;2. PMID 8959493
- [Background] Cejna M, Thurnher S, Illiasch H, Horvath W, Waldenberger P, Hornik K, Lammer J. PTA versus Palmaz stent placement in femoropopliteal artery obstructions: a multicenter prospective randomized study. J Vasc Interv Radiol. 2001 Jan;12(1):23-31. doi: 10.1016/s1051-0443(07)61397-9. PMID 11200349
- [Background] Vroegindeweij D, Vos LD, Tielbeek AV, Buth J, vd Bosch HC. Balloon angioplasty combined with primary stenting versus balloon angioplasty alone in femoropopliteal obstructions: A comparative randomized study. Cardiovasc Intervent Radiol. 1997 Nov-Dec;20(6):420-5. doi: 10.1007/s002709900186. PMID 9354709
- [Background] Grimm J, Muller-Hulsbeck S, Jahnke T, Hilbert C, Brossmann J, Heller M. Randomized study to compare PTA alone versus PTA with Palmaz stent placement for femoropopliteal lesions. J Vasc Interv Radiol. 2001 Aug;12(8):935-42. doi: 10.1016/s1051-0443(07)61572-3. PMID 11487673
- [Background] Zdanowski Z, Albrechtsson U, Lundin A, Jonung T, Ribbe E, Thorne J, Norgren L. Percutaneous transluminal angioplasty with or without stenting for femoropopliteal occlusions? A randomized controlled study. Int Angiol. 1999 Dec;18(4):251-5. PMID 10811511
- [Background] Becquemin JP, Favre JP, Marzelle J, Nemoz C, Corsin C, Leizorovicz A. Systematic versus selective stent placement after superficial femoral artery balloon angioplasty: a multicenter prospective randomized study. J Vasc Surg. 2003 Mar;37(3):487-94. doi: 10.1067/mva.2003.155. PMID 12618680
- [Background] Schillinger M, Minar E. Endovascular stent implantation for treatment of peripheral artery disease. Eur J Clin Invest. 2007 Mar;37(3):165-70. doi: 10.1111/j.1365-2362.2007.01774.x. PMID 17359483
- [Background] Tetteroo E, van der Graaf Y, Bosch JL, van Engelen AD, Hunink MG, Eikelboom BC, Mali WP. Randomised comparison of primary stent placement versus primary angioplasty followed by selective stent placement in patients with iliac-artery occlusive disease. Dutch Iliac Stent Trial Study Group. Lancet. 1998 Apr 18;351(9110):1153-9. doi: 10.1016/s0140-6736(97)09508-1. PMID 9643685